CLINICAL TRIAL: NCT03420157
Title: Carrying Out of Focus Group to Improve Cervical Screening Proposal by Vaginal Self-sampling (APACHE-4/FG).
Acronym: APACHE-4/FG
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: INCA17-JB/APACHE-4/FG
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Cancer Cervix
Keywords: Cervical cancer screening; vaginal self-sampling; Focus group; communication
MeSH Terms: conditions — Uterine Cervical Neoplasms; Communication | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus Group 1 & 2: Each Focus Group of 10 women will be led by a psychologist according to a semi-directive interview pattern. This interview guideline specifies in details the ideal proceedings of Focus Group, as well as the various predetermined topics to be addressed in the form of questions and / or relaunches. The interview guideline is divided into 2 parts: the accompanying letter and the leaflet explaining how to perform the vaginal self-sampling.
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: Focus Group — Focus Group of 2 hours. Women will be asked to give their opinion about the communication media of the vaginal self-sampling kit.

SUMMARY:
Despite the existence of an effective screening test (pap smear), cervical cancer is, every year in France, the cause of more than 3,000 new cases and 1,100 deaths. But, in France, 4 in 10 women are not screened or not often enough (nearly 7 millions women). It is therefore necessary to develop new strategies to reach these women. The etiological factor of this cancer is persistent infection with oncogenic High-Risk Human PapillomaVirus (HR-HPV). Thereby, HPV-based tests could be alternative screening tests. Vaginal self-sampling with HR-HPV test is simpler and less intrusive than the pap smear. It has been shown that vaginal self-sampling with HPV test is a powerful means to increase the participation rate in cervical cancer screening. The investigators hypothesize that it is possible to optimize participation rate by improving the communication media associated to the vaginal self-sampling kit. This is why the accompanying letter and the leaflet explaining how to perform the vaginal self-sampling will be submit to women opinion by using the Focus Group method. The objective is to identify improvement ideas of these two communication media.

ELIGIBILITY:
Inclusion Criteria:

* women from 30 to 65 years old
* women living in french territorial division 37 ("Indre-et-Loire")
* no pap smear made in the three last years (ideally)

Exclusion Criteria:

* Follow-up in progress for positive screening

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty women living near the city of Tours not screened by pap smear (ideally since at least 3 years). Women who could be interested by the vaginal self-sampling screening alternative.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2018-02-08 (Actual)

PRIMARY OUTCOMES:
Focus group methodology (structured questionnaire) will use to identify group norms or a range of views and to capitalise on the interaction within the group to identify levers and brakes and improve communication media (10 women for each focus group) | A systematic text analysis of the transcripts will be performed after data saturation was reached (projection: 2 focus group of 2 hours in two weeks)
  The transcripts of the discussions will be reviewed by the psychologist to identify the emerging themes (anxiety, motivating information, ...) to identify levers and brakes and improve communication media.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Boyard, Principal Investigator — Centre de coordination des dépistages des cancers, CHRU de Tours
Locations (1):
- UH Tours, Tours, Indre-et-Loire, France